CLINICAL TRIAL: NCT03351920
Title: Ventilation's Parameters Applied in Emergency Medicine. Observational Study
Brief Title: Ventilation's Parameters Applied in Emergency Medicine. A Prospective Observational Study
Acronym: PARAVENT
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PARAVENT
Record Dates: First submitted 2017-10-24; First posted 2017-11-24 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Mechanical Ventilation; Acute Respiratory Distress Syndrome; Protective Ventilation; Survival
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: mechanical ventilation — All patients who need an invasive or non invasive mechanical ventilation, initiated in Prehospital or IntraHospital Emergency Department by an emergency Physician

SUMMARY:
To prospectively assess the mechanical ventilation management when its provided by Emergency Physicians in French Hospital, and to assess complications and outcome of these patients.

The study could be measure the proportion of patients developing an Acute Respiratory Failure Distress after a take care of by French Emergency Departments.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or over 18 years old
* Needing a invasive or noninvasive mechanical ventilation
* Mechanical ventilation initiated in Prehospital or IntraHospital Emergency Department by an Emergency Physician

Exclusion Criteria:

- Age under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who need an invasive or non invasive mechanical ventilation, initiated in Prehospital or IntraHospital Emergency Department by an emergency Physician
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients benefiting of a early low-volume ventilation initiated Emergency Department or Prehospital Care. | Day 1
  Early Low volume ventilation will be defined according to a VtE < 8mL/lg

SECONDARY OUTCOMES:
Proportion of patients benefiting of an early protective ventilation in Emergency Departments | Day 1
Proportion of patients with acute respiratory distress syndrome according to the Berlin Definition during the first eight days of following. | from Day 1 to Day 8 and Day 28
  ARDS will be defined according to the Berlin definition.
Proportion of survival from day 1 to Day 8, and to day 28 | from Day 1 to Day 8 and Day 28
Indication to mechanical ventilation in Prehospital care and Emergency Departments | Day 1
Mechanical Ventilation Duration in Emergency Departments | Day 1
Mechanical ventilation settings in Emergency Departments | Day 1
  Recorded settings will be Ventilation mode, Tidal volume or Pressure Support Positive End Expiratory Pressure, Ventilation Rate, I : E ratio or Inspiratory Flow or Inspiratory Time.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Pierre-Arnaud Fort, Agen
  - CHU de Bordeaux, Bordeaux
  - Pierre-Marie Noël, Brest
  - Paul Fievet, La Rochelle
  - Thomas Lenormand, Lorient
  - CH de Niort, Niort
  - Marjanovic Nicolas, Poitiers